CLINICAL TRIAL: NCT05003739
Title: A Post-market Study Evaluating Clinical and Radiographic Early Outcomes of Hip Arthroplasty With Logica Mirror Stem.
Brief Title: Hip Arthroplasty With Logica Mirror Femoral Stem
Status: Active, not recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-37
Record Dates: First submitted 2021-07-19; First posted 2021-08-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hip Replacement
Keywords: Cemented femoral stem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Logica Mirror: Since the trial is not comparative, the only arm implies the use of the investigational device (Logica Mirror femoral stem)
  Interventions: Procedure: Hip arthroplasty with Logica Mirror femoral stem

INTERVENTIONS:
Procedure: Hip arthroplasty with Logica Mirror femoral stem — Total or partial hip arthroplasty with implant of Logica Mirror femoral stem

SUMMARY:
Logica Mirror femoral stem is a CE marked medical device, and within this clinical trial it is used according to its intended use. This is a Post Marketing Clinical Follow Up trial, with the main aim to collect additional evidences on the outcome data on this product, by analysing clinical scoring systems, radiographs and adverse event records within three years after the surgery, and thus to assess the short-term performance and safety of this implant.

ELIGIBILITY:
All patients that underwent partial or total hip arthroplasty and implanted with LOGICA MIRROR femoral stem between Jan 2010 and Dec 2021 at Nemocnice Kyjov Hospital (CZ) in accordance with the indication for use of the product and site standard of practice.

Additional Inclusion criteria:

* Availability of patients' immediate post-operative radiograph (baseline) and of a number of follow-up x-rays that the Principal Investigator deems sufficient for an effective radiographic implant evaluation and stability assessment;
* Patient is willing and able to complete additional follow-up evaluations if needed after signing ICF.

Exclusion criteria

* Age < 18 years;
* Female patients who are pregnant, nursing, or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Nemocnice Kyjov Hospital (CZ)
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score - Functional change | From preoperative (baseline) to 3 years after surgery
  Functional change in Harris Hip Score (HHS). The maximum score of HHS is 100 points. Pain domain contributes 44 points, function 47, ROM 5 and absence of deformity 4 points.
  Results can be interpreted with the following: Less than 60= failed result; 60 to 69= poor result; 70 to 79= fair; 80 to 90= good; 90 to 100= excellent;

SECONDARY OUTCOMES:
Oxford Hip Score - Functional change | From preoperative (baseline) to 3 years after surgery
  Functional change in Oxford Hip Score. The OHS is a short 12-item survey. It comprises two domains (pain and function), with six items or questions in each, using the following scoring: each question has been scored between 0 and 4, with 4 being the best outcome, producing overall scores running from 0 to 48, with 48 being the best outcome.
  The calculation of the total score of OHS is based on this scoring system and the resulted score can be interpreted as follows: less than 27 points= poor; 27 to 33 points= fair; 34 to 41 points= good; 41 to 48 points= excellent
VAS satisfaction | From 6 weeks to 3 years after surgery
  Functional evaluation of VAS satisfaction.
  Patient is asked to rate his satisfaction by making a vertical mark on the 100-mm line. The measurement in millimetres is eventually converted to the same number of points ranging from 0 to 100 points
Radiographic implant evaluation and stability assessment of Logica Mirror stem | From discharge to 3 years after surgery
  Stability assessment of Logica Mirror stem (through radiographic implant evaluation).
  For assessing the stability of the femoral component in a cemented configuration, the presence of radiolucent lines should be recorded both at stem-cement interface and at cement-bone interface.
  At each postoperative time-point the radiolucencies will be measured in every Gruen zone and graded in accordance to the following classification:
  None: No evidence of radiolucency
  1. mm: Presence of 1 mm-width radiolucent lines
  2. mm: Presence of 2 mm-width radiolucent lines > 2 mm: Presence of radiolucent lines wider than 2 mm
Survival rate of the implant | 3 years
  Survival rate of the implant (Kaplan-Meier) at 3 years after surgery
Safety profile of Logica Mirror by recording adverse events (AE), serious adverse events (SAE), device deficiency (DD), adverse device effect (ADE), serious adverse device effect (SADE) | From intraoperative to 3 years after surgery
  Incidence of device-related adverse events( AE), serious adverse events (SAE), device deficiency (DD), adverse device effect (ADE), serious adverse device effect (SADE).

CONTACTS AND LOCATIONS:
Locations (1):
- Nemocnice Kyjov Hospital, Kyjov, CZ Republic, Czechia

IPD SHARING:
Plan to Share IPD: No